CLINICAL TRIAL: NCT03555591
Title: Specified Drug-Use Survey of Trelagliptin Tablets "Survey on Long-term Use in Patients With Type 2 Diabetes Mellitus"
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: Trelagliptin-5001; JapicCTI-183980 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2018-06-01; First posted 2018-06-13 (Actual); Results first posted 2023-09-01 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — trelagliptin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Trelagliptin 100 mg: Trelagliptin 100 mg tablet, orally, once weekly for up to 36 months. Participants received interventions as part of routine medical care.
  Interventions: Drug: Trelagliptin

INTERVENTIONS:
Drug: Trelagliptin — Trelagliptin tablets
  Other Names: Zafatek tablets

SUMMARY:
The purpose of this survey is to evaluate the long-term safety and efficacy of trelagliptin tablets in patients with type 2 diabetes mellitus in the routine clinical setting.

DETAILED DESCRIPTION:
The drug being tested in this survey is called trelagliptin tablet. This tablet is being tested to treat people who have type 2 diabetes mellitus.

This survey is an observational (non-interventional) study and will look at the long-term safety and efficacy of the trelagliptin tablet in the routine clinical setting. The planned number of observed patients will be approximately 3000.

This multi-center observational trial will be conducted in Japan.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus patients

Exclusion Criteria:

1. Have severe ketosis, diabetic coma or precoma, or type 1 diabetes mellitus
2. Have severe infection, perioperative status, or serious trauma
3. Have severe renal impairment or on dialysis due to end-stage renal disease
4. Have a history of hypersensitivity to any ingredients of this drug

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with type 2 diabetes mellitus in the routine clinical setting
Sampling Method: Probability Sample
Enrollment: 3198 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Takeda Selected Site, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5f6b60394db2bf003ab4a1de

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the survey at 242 investigative sites in Japan, from 1 May 2016 to 31 October 2021.
Pre-assignment Details: Participants with a historical diagnosis of type 2 diabetes mellitus were enrolled. Participants received trelagliptin as part of a routine medical care.
Period: Overall Study
Arm/Group | Trelagliptin 100 mg
Started | 3198
Completed | 3121
Not Completed | 77
Not completed — Protocol Violation | 77

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set, The safety analysis set was defined as all participants who completed the survey.
Arm/Group | Trelagliptin 100 mg
Number analyzed (Participants) | 3121
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.8 (12.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1870
  Male | 1251
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants] — All participants were enrolled in Japan.
  Participants
    Japan | 3121
Duration of Type 2 Diabetes Mellitus [Mean (Standard Deviation); unit: Years] — Mean duration between the first diagnosis of type 2 diabetes mellitus and the start of the study was reported. Population: The number analyzed is the number of participants with data available for analysis.
  Years
    number analyzed (Participants) | 2068
    (all) | 7.6 (7.28)
Weight [Mean (Standard Deviation); unit: Kilogram (kg)] — Population: The number analyzed is the number of participants with data available for analysis.
  Kilogram (kg)
    number analyzed (Participants) | 2183
    (all) | 65.12 (14.293)
BMI [Mean (Standard Deviation); unit: Kilogram (kg)/meter (m)^2] — Body Mass Index = weight (kg)/[height (m)^2] Population: The number analyzed is the number of participants with data available for analysis.
  Kilogram (kg)/meter (m)^2
    number analyzed (Participants) | 2006
    (all) | 24.94 (4.217)
Height [Mean (Standard Deviation); unit: Centimeters (cm)] — Population: The number analyzed is the number of participants with data available for analysis.
  Centimeters (cm)
    number analyzed (Participants) | 2396
    (all) | 161.1 (9.95)
Healthcare Category [Count of Participants; unit: Participants] — Participants were categorized as outpatient and inpatient.
  Participants
    Outpatient | 3081
    Inpatient | 40
Predisposition to Hypersensitivity [Count of Participants; unit: Participants] — Number of participants who had or did not have a liability or tendency to suffer from hypersensitivity was reported. Unknown: Data could not be collected.
  Participants
    Had No Predisposition to Hypersensitivity | 2744
    Had Predisposition to Hypersensitivity | 144
    Unknown | 233
Medical Complications [Count of Participants; unit: Participants] — Complications defined as a disease or a health condition for each participant at the start of study. Complications were classified as congenital anomalies, endocrine disorders, hematologic disorders, psychiatric and nervous system disorders, cardiovascular disorders, respiratory disorders, gastrointestinal (GI) disorders, renal disease and other complications. Other complications included all complications except for those mentioned above.
  Participants
    Had No Medical Complications | 609
    Had Medical Complications | 2512
Medical History [Count of Participants; unit: Participants] — Medical history defined as a disease or a health condition for each participant before start of the study. Medical history was classified as congenital anomalies, hematologic disorders, psychiatric and nervous system disorders, cardiovascular disorders, respiratory disorders, GI disorders, hepatic and biliary disorders, renal disease and other medical history. Other medical history included all medical history except for those mentioned above. Unknown: Data could not be collected.
  Participants
    Had No Medical History | 2383
    Had Medical History | 500
    Unknown | 238
Smoking Classification [Count of Participants; unit: Participants] — Unknown: Data could not be collected.
  Participants
    Never Smoked | 1407
    Current Smoker | 391
    Ex-Smoker | 637
    Unknown | 686
Alcohol Classification [Count of Participants; unit: Participants] — Participants who answered Yes or No for a question "Drink Alcohol Almost Every Day?" were reported. Unknown: Data could not be collected.
  Participants
    Yes | 645
    No | 1863
    Unknown | 613
Renal Impairment [Count of Participants; unit: Participants]
  Had No Renal Impairment | 2739
  Had Renal Impairment | 382
Hepatic Impairment [Count of Participants; unit: Participants]
  Had No Hepatic Impairment | 2578
  Had Hepatic Impairment | 543
Glycosylated Hemoglobin A1c (HbA1c) [National Glycohemoglobin Standardization Program (NGSP)] [Mean (Standard Deviation); unit: Percent] — Population: The number analyzed is the number of participants with data available for analysis.
  Percent
    number analyzed (Participants) | 2635
    (all) | 7.38880 (1.348643)
Fasting Blood Glucose [Mean (Standard Deviation); unit: milligram (mg)/deciliter (dL)] — Population: The number analyzed is the number of participants with data available for analysis.
  milligram (mg)/deciliter (dL)
    number analyzed (Participants) | 1494
    (all) | 151.379 (59.8728)
Fasting Glucagon [Mean (Standard Deviation); unit: picogram (pg)/milliliter (mL)] — Population: The number analyzed is the number of participants with data available for analysis.
  picogram (pg)/milliliter (mL)
    number analyzed (Participants) | 83
    (all) | 177.52 (55.766)
Serum Creatinine Value Within 1 Month Before Start of Treatment with the Study Drug [Mean (Standard Deviation); unit: mg/dL] — Population: The number analyzed is the number of participants with data available for analysis.
  mg/dL
    number analyzed (Participants) | 2778
    (all) | 0.7717 (0.21925)
Creatinine Clearance Within 1 Month Before Start of Treatment with the Study Drug [Mean (Standard Deviation); unit: mL/minute (min)] — Population: The number analyzed is the number of participants with data available for analysis.
  mL/minute (min)
    number analyzed (Participants) | 1922
    (all) | 89.54 (41.618)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Had One or More Adverse Events
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment.
Time Frame: 36 months
Population: Safety Analysis Set, The safety analysis set was defined as all participants who completed the survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Trelagliptin 100 mg
Number analyzed (Participants) | 3121
Participants | 390

2. Primary Outcome: Number of Participants Who Had One or More Adverse Drug Reactions
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. Adverse drug reaction refers to AE related to administered drug.
Time Frame: 36 months
Population: Safety Analysis Set, The safety analysis set was defined as all participants who completed the survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Trelagliptin 100 mg
Number analyzed (Participants) | 3121
Participants | 96

3. Secondary Outcome: Change From Baseline in Mean Glycosylated Hemoglobin (HbA1c)
Description: The reported data was the change in the mean value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected between baseline and timepoints (up to final assessment point: Month 36). A negative change from baseline indicates improvement.
Time Frame: Baseline, up to final assessment point (up to Month 36)
Population: Efficacy assessment population, The efficacy assessment population was defined as participants who completed the survey and had efficacy data at baseline and post-baseline time points available.
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Trelagliptin 100 mg
Number analyzed (Participants) | 3121
Percent
  Month 1: number analyzed (Participants) | 1795
  Month 1 | -0.24813 (0.682526)
  Month 3: number analyzed (Participants) | 2161
  Month 3 | -0.40573 (1.136176)
  Month 6: number analyzed (Participants) | 2190
  Month 6 | -0.43716 (1.173372)
  Month 12: number analyzed (Participants) | 2153
  Month 12 | -0.44281 (1.131737)
  Month 18: number analyzed (Participants) | 1820
  Month 18 | -0.33933 (1.181299)
  Month 24: number analyzed (Participants) | 1723
  Month 24 | -0.34909 (1.194628)
  Month 30: number analyzed (Participants) | 1564
  Month 30 | -0.33164 (1.194041)
  Month 36: number analyzed (Participants) | 1540
  Month 36 | -0.35018 (1.197507)
  Final Assessment Point (Up to Month 36): number analyzed (Participants) | 2583
  Final Assessment Point (Up to Month 36) | -0.33498 (1.328413)

4. Secondary Outcome: Change From Baseline in Fasting Blood Glucose
Description: The reported data was the change in the mean value of fasting blood glucose collected between baseline and timepoints (up to final assessment point: Month 36). A negative change from baseline indicates improvement.
Time Frame: Baseline, up to final assessment point (up to Month 36)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Trelagliptin 100 mg
Number analyzed (Participants) | 3121
mg/dL
  Month 1: number analyzed (Participants) | 837
  Month 1 | -11.733 (50.2247)
  Month 3: number analyzed (Participants) | 1073
  Month 3 | -11.896 (50.4982)
  Month 6: number analyzed (Participants) | 1106
  Month 6 | -13.816 (57.8209)
  Month 12: number analyzed (Participants) | 1130
  Month 12 | -14.698 (53.3678)
  Month 18: number analyzed (Participants) | 813
  Month 18 | -10.999 (55.6319)
  Month 24: number analyzed (Participants) | 778
  Month 24 | -7.056 (58.7981)
  Month 30: number analyzed (Participants) | 716
  Month 30 | -9.183 (58.2264)
  Month 36: number analyzed (Participants) | 711
  Month 36 | -9.928 (55.3334)
  Final Assessment Point (Up to Month 36): number analyzed (Participants) | 1417
  Final Assessment Point (Up to Month 36) | -9.765 (59.2496)

5. Secondary Outcome: Change From Baseline in Fasting Insulin Level
Description: The reported data was the change in the mean value of fasting insulin level collected between baseline and timepoints (up to final assessment point: Month 36).
Time Frame: Baseline, up to final assessment point (up to Month 36)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: microunit/milliliter (mcrU/mL)
Arm/Group | Trelagliptin 100 mg
Number analyzed (Participants) | 3121
microunit/milliliter (mcrU/mL)
  Month 1: number analyzed (Participants) | 71
  Month 1 | -7.079 (19.5631)
  Month 3: number analyzed (Participants) | 93
  Month 3 | -5.520 (19.7015)
  Month 6: number analyzed (Participants) | 96
  Month 6 | -6.999 (18.9998)
  Month 12: number analyzed (Participants) | 112
  Month 12 | -4.354 (18.4697)
  Month 18: number analyzed (Participants) | 93
  Month 18 | -4.905 (15.3859)
  Month 24: number analyzed (Participants) | 83
  Month 24 | -6.601 (16.6195)
  Month 30: number analyzed (Participants) | 78
  Month 30 | -7.114 (17.3951)
  Month 36: number analyzed (Participants) | 68
  Month 36 | -5.740 (18.2392)
  Final Assessment Point (Up to Month 36): number analyzed (Participants) | 129
  Final Assessment Point (Up to Month 36) | -4.675 (15.9822)

6. Secondary Outcome: Change From Baseline in Homeostasis Model Assessment of Beat-cell Function (HOMA-beta)
Description: The reported data was the change in the mean value of HOMA-beta. HOMA-beta measures as following; HOMA-beta = fasting insulin (microU/mL) ×360/ [fasting glucose (mg/dL) - 63].
Time Frame: Baseline, up to final assessment point (up to Month 36)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Trelagliptin 100 mg
Number analyzed (Participants) | 3121
Percent
  Month 1: number analyzed (Participants) | 71
  Month 1 | -26.523 (106.9238)
  Month 3: number analyzed (Participants) | 91
  Month 3 | -21.155 (116.4317)
  Month 6: number analyzed (Participants) | 96
  Month 6 | -23.442 (107.4707)
  Month 12: number analyzed (Participants) | 111
  Month 12 | -16.312 (104.6056)
  Month 18: number analyzed (Participants) | 93
  Month 18 | -21.949 (104.5351)
  Month 24: number analyzed (Participants) | 83
  Month 24 | -34.083 (102.0591)
  Month 30: number analyzed (Participants) | 78
  Month 30 | -39.639 (120.4540)
  Month 36: number analyzed (Participants) | 68
  Month 36 | -31.484 (129.2697)
  Final Assessment Point (Up to Month 36): number analyzed (Participants) | 128
  Final Assessment Point (Up to Month 36) | -19.551 (106.4136)

7. Secondary Outcome: Change From Baseline in Fasting Glucagon
Description: The reported data was the change in the mean value of fasting glucagon collected between baseline and timepoints (up to final assessment point: Month 36).
Time Frame: Baseline, up to final assessment point (up to Month 36)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Trelagliptin 100 mg
Number analyzed (Participants) | 3121
pg/mL
  Month 1: number analyzed (Participants) | 67
  Month 1 | -7.88 (46.589)
  Month 3: number analyzed (Participants) | 74
  Month 3 | -9.22 (51.995)
  Month 6: number analyzed (Participants) | 72
  Month 6 | 6.65 (42.295)
  Month 12: number analyzed (Participants) | 73
  Month 12 | -1.41 (46.540)
  Month 18: number analyzed (Participants) | 67
  Month 18 | 10.38 (51.088)
  Month 24: number analyzed (Participants) | 61
  Month 24 | -3.56 (54.207)
  Month 30: number analyzed (Participants) | 37
  Month 30 | 18.65 (91.492)
  Month 36: number analyzed (Participants) | 46
  Month 36 | 0.18 (82.427)
  Final Assessment Point (Month 36): number analyzed (Participants) | 81
  Final Assessment Point (Month 36) | 4.27 (70.248)

8. Secondary Outcome: Percentage of Participants Achieving Good Glycemic Control (Reduction in HbA1c Values < 8.0 Percent)
Description: The reported data was percentage of participants who achieved good glycemic control (defined as reduction in HbA1c values < 8.0 Percent) at baseline and timepoints (up to final assessment point: Month 36).
Time Frame: Baseline, up to final assessment point (up to Month 36)
Population: as for outcome 3
Measure: Number; unit: Percent
Arm/Group | Trelagliptin 100 mg
Number analyzed (Participants) | 3121
Percent
  Baseline: number analyzed (Participants) | 2635
  Baseline | 78.0
  Month 1: number analyzed (Participants) | 2045
  Month 1 | 81.9
  Month 3: number analyzed (Participants) | 2411
  Month 3 | 86.1
  Month 6: number analyzed (Participants) | 2491
  Month 6 | 87.3
  Month 12: number analyzed (Participants) | 2502
  Month 12 | 88.8
  Month 18: number analyzed (Participants) | 2054
  Month 18 | 87.5
  Month 24: number analyzed (Participants) | 1947
  Month 24 | 88.1
  Month 30: number analyzed (Participants) | 1784
  Month 30 | 88.4
  Month 36: number analyzed (Participants) | 1822
  Month 36 | 89.3
  Final Assessment Point (Up to Month 36): number analyzed (Participants) | 3046
  Final Assessment Point (Up to Month 36) | 84.6

9. Secondary Outcome: Percentage of Participants Achieving Good Glycemic Control (Reduction in HbA1c Values < 7.0 Percent)
Description: The reported data was percentage of participants who achieved good glycemic control (defined as reduction in HbA1c values < 7.0 Percent) at baseline and timepoints (up to final assessment point: Month 36).
Time Frame: Baseline, up to final assessment point (up to Month 36)
Population: as for outcome 3
Measure: Number; unit: Percent
Arm/Group | Trelagliptin 100 mg
Number analyzed (Participants) | 3121
Percent
  Baseline: number analyzed (Participants) | 2635
  Baseline | 44.3
  Month 1: number analyzed (Participants) | 2045
  Month 1 | 50.3
  Month 3: number analyzed (Participants) | 2411
  Month 3 | 58.4
  Month 6: number analyzed (Participants) | 2491
  Month 6 | 60.9
  Month 12: number analyzed (Participants) | 2502
  Month 12 | 62.5
  Month 18: number analyzed (Participants) | 2054
  Month 18 | 58.5
  Month 24: number analyzed (Participants) | 1947
  Month 24 | 60.0
  Month 30: number analyzed (Participants) | 1784
  Month 30 | 59.7
  Month 36: number analyzed (Participants) | 1822
  Month 36 | 63.1
  Final Assessment Point (Up to Month 36): number analyzed (Participants) | 3046
  Final Assessment Point (Up to Month 36) | 58.0

10. Secondary Outcome: Percentage of Participants Achieving Good Glycemic Control (Reduction in HbA1c Values < 6.0 Percent)
Description: The reported data was percentage of participants who achieved good glycemic control (defined as reduction in HbA1c values < 6.0 Percent) at baseline and timepoints (up to final assessment point: Month 36).
Time Frame: Baseline, up to final assessment point (up to Month 36)
Population: as for outcome 3
Measure: Number; unit: Percent
Arm/Group | Trelagliptin 100 mg
Number analyzed (Participants) | 3121
Percent
  Baseline: number analyzed (Participants) | 2635
  Baseline | 6.0
  Month 1: number analyzed (Participants) | 2045
  Month 1 | 6.8
  Month 3: number analyzed (Participants) | 2411
  Month 3 | 8.7
  Month 6: number analyzed (Participants) | 2491
  Month 6 | 9.8
  Month 12: number analyzed (Participants) | 2502
  Month 12 | 11.0
  Month 18: number analyzed (Participants) | 2504
  Month 18 | 8.2
  Month 24: number analyzed (Participants) | 1947
  Month 24 | 8.1
  Month 30: number analyzed (Participants) | 1784
  Month 30 | 9.3
  Month 36: number analyzed (Participants) | 1822
  Month 36 | 11.2
  Final Assessment Point (Up to Month 36): number analyzed (Participants) | 3046
  Final Assessment Point (Up to Month 36) | 11.3

ADVERSE EVENTS:
Time Frame: 36 months
Description: At each visit the investigator had to document any occurrence of AEs and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to the survey treatment.
Arm/Group | Trelagliptin 100 mg
All-Cause Mortality (participants affected / at risk) | 24/3121
Serious Adverse Events (participants affected / at risk) | 167/3121
Other Adverse Events (participants affected / at risk) | 54/3121
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trelagliptin 100 mg (N=3121)
Cellulitis (Infections and infestations) | 2
Diabetic gangrene (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Liver abscess (Infections and infestations) | 1
Meningitis aseptic (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 5
Pneumonia aspiration (Infections and infestations) | 2
Pneumonia pneumococcal (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Pyelonephritis acute (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 2
Hepatitis B reactivation (Infections and infestations) | 1
Bacterial pyelonephritis (Infections and infestations) | 1
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Biliary neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Carcinoid tumour of the gastrointestinal tract (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Anaemia (Blood and lymphatic system disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 1
Thrombocytopenic purpura (Blood and lymphatic system disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 15
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 8
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1
Ketoacidosis (Metabolism and nutrition disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1
Completed suicide (Psychiatric disorders) | 1
Schizophrenia (Psychiatric disorders) | 1
Altered state of consciousness (Nervous system disorders) | 1
Cerebral infarction (Nervous system disorders) | 6
Embolic stroke (Nervous system disorders) | 1
Facial paralysis (Nervous system disorders) | 1
Neuropathy peripheral (Nervous system disorders) | 1
Subarachnoid haemorrhage (Nervous system disorders) | 1
Metabolic encephalopathy (Nervous system disorders) | 1
Carotid arteriosclerosis (Nervous system disorders) | 3
Cataract nuclear (Eye disorders) | 1
Retinopathy (Eye disorders) | 1
Sudden hearing loss (Ear and labyrinth disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 1
Angina pectoris (Cardiac disorders) | 5
Angina unstable (Cardiac disorders) | 1
Arrhythmia (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 4
Atrioventricular block complete (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 2
Cardiac tamponade (Cardiac disorders) | 1
Coronary artery stenosis (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Myocardial ischaemia (Cardiac disorders) | 2
Ventricular extrasystoles (Cardiac disorders) | 1
Acute coronary syndrome (Cardiac disorders) | 1
Peripheral artery occlusion (Vascular disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Idiopathic interstitial pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2
Mechanical ileus (Gastrointestinal disorders) | 1
Large intestine polyp (Gastrointestinal disorders) | 1
Autoimmune pancreatitis (Gastrointestinal disorders) | 2
Autoimmune hepatitis (Hepatobiliary disorders) | 1
Bile duct stone (Hepatobiliary disorders) | 1
Cholangitis acute (Hepatobiliary disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 2
Chronic hepatitis (Hepatobiliary disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 1
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Postrenal failure (Renal and urinary disorders) | 1
Renal impairment (Renal and urinary disorders) | 5
Chronic kidney disease (Renal and urinary disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Ureterolithiasis (Renal and urinary disorders) | 1
Ovarian cyst (Reproductive system and breast disorders) | 1
Oedema peripheral (General disorders) | 1
Sudden death (General disorders) | 1 — The reasons of events are not determined because assessment findings were insufficient to specify the reason.
Multiple organ dysfunction syndrome (General disorders) | 1
Electrocardiogram QT prolonged (Investigations) | 1
Electrocardiogram Q wave abnormal (Investigations) | 1
Blood alkaline phosphatase increased (Investigations) | 1
Hepatic enzyme increased (Investigations) | 1
Patella fracture (Injury, poisoning and procedural complications) | 1
Rib fracture (Injury, poisoning and procedural complications) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1
Transcatheter aortic valve implantation (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Trelagliptin 100 mg (N=3121)
Hypertension (Vascular disorders) | 54

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2020-12-25): https://cdn.clinicaltrials.gov/large-docs/91/NCT03555591/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-07): https://cdn.clinicaltrials.gov/large-docs/91/NCT03555591/SAP_001.pdf